CLINICAL TRIAL: NCT06855680
Title: The EMIRATES Study - Development and Evaluation of Thyroid Cancer Patient Decision Aid (PDA-TC) - Pilot Study
Brief Title: The EMIRATES Study
Status: Recruiting | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Wrightington, Wigan and Leigh NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR5869
Record Dates: First submitted 2024-10-03; First posted 2025-03-04 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2024-10

CONDITIONS: Differentiated Thyroid Cancer (DTC)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control arm: Control arm will follow standard clinical practice. Patients with newly diagnosed low-risk DTC will be recruited to attend two outpatient clinical appointments as part of their standard thyroid cancer care pathway. In the initial consultation, thyroid cancer clinicians will discuss with patient the available treatment options (i.e. total thyroidectomy and hemithyroidectomy) for the low-risk DTC and their associated risks and benefits. Instead of making the treatment decision straight away, patients will be allowed to a week to digest the information and to consider the options. A week later, patients will return for the second outpatient consultation where they will decide on the treatment with their clinicians.
- PDA arm: In the PDA arm, the study procedure will be the same as in control arm except that the PDA-TC pamphlet will be introduced to patient after the first outpatient clinical consultation. Patients are allowed to take the PDA-TC home to read and digest the information before returning for their second outpatient consultation a week later. The data collection timing and measures in the PDA arm will remain the same as in the control arm.

SUMMARY:
This pilot study will take place in thyroid outpatient clinics. It will have two study arms running in consecutive order: first, a Control arm where standard care will take place without PDA-TC, then a Patient Decision Aid (PDA) arm where the PDA-TC is implemented into the clinical practice. Within each arm, eligible patients will attend two thyroid cancer outpatient clinical consultations during which the patient will make a shared decision with their clinicians regarding surgical treatment between hemithyroidectomy and total thyroidectomy. In the PDA arm, the PDA TC pamphlet will be introduced to study participants after the initial clinical consultation. The participants will be encouraged to read and digest information related to the disease and treatment options on PDA-TC before returning for their second consultation where a treatment decision will be made together with their clinicians. Participants will be asked to complete the Decisional Conflict Scale questionnaire after each consultation in both study arms. The patient will also complete a Satisfaction with Decision Scale questionnaire and a Preparation for Decision Making Scale questionnaire after the second consultation in both arms.

DETAILED DESCRIPTION:
PDA-TC is an education pamphlet which helps patient become involved in decision-making by providing information about the treatment options and their outcomes and by clarifying personal values. This pilot study of PDA-TC will involve a cross-sectional prospective observational pilot study.

The thyroid cancer incidence rates have increased by more than two-and-half times (175%) in the UK since early 1990s. The surge of differentiated thyroid cancer (DTC) has been suggested to be at least partly owing to overdiagnosis. Due to the widespread use of advanced imaging and increased pathological scrutiny of thyroid specimens, the majority of these cases are small/early low-risk cancers. Around 72% of thyroid cancer cases in the UK are in females and the disease is often diagnosed at a younger age (30 to 50), compared to other adult cancers. Until 2015, the standard of care for DTC has been a 'one size fits all' approach of total thyroidectomy (TT) for more than 1 cm DTC which may be followed with adjuvant radioactive iodine ablation. This treatment has afforded excellent overall survival rate (98-99% at 10-year) and a low recurrence rate (2-8% at 7-year). However, this survival benefit comes at the price of life-long hormone replacement therapy and increased risk of post-operative complication such as vocal cord paralysis and hypoparathyroidism. These negative ramifications of TT have a huge implication on thyroid patient's physical and emotional functioning, their working and family life, and long-term quality of life (QoL).

In addition, a significant number of DTC cannot be confirmed with needle biopsy. Therefore, TT is often performed in two stages with diagnostic hemithyroidectomy (HT) of the main lobe first (to confirm the diagnosis) while the remain gland is excised at a later stage, subjecting patient to two operations. In response to widely published concerns about overdiagnosis and overtreatment, both the British Thyroid Association 2014 guideline and the American Thyroid Association 2015 guideline have endorsed hemithyroidectomy (HT) as an alternative treatment approach to TT for DTC. This is because TT does not appear to offer an overall survival advantage over HT. Although HT is generally better tolerated by patient, it carries a higher cancer recurrence rate when compared with TT. In the UK, many thyroid cancer multidisciplinary teams and surgeons have started to offer HT to low-risk DTC patients while other centres continue to recommend TT as the main treatment approach. A clear clinical equipoise therefore exists for managing low-risk thyroid cancer. When faced with this equipoise, where clinicians are not sure and data are still equivocal, it is even more difficult for patients to understand the issues and make a treatment choice that is best for their individual needs and priorities. Due to the excellent prognosis, there is an ever-increasing pool of cancer-survivors in whom maintaining a good long-term QoL has become an integral part of their cancer care. Unfortunately, studies have shown that thyroid cancer survivors have a reduced QoL that is similar to or worse than those with more aggressive malignancies, such as breast or colon cancer. A recent National Patient Survey showed that the existing clinical equipoise has resulted in high level of confusion, dissatisfaction, and anxiety in patients with regards to treatment decision.

Shared Decision Making (SDM) is characterised by intentional and cooperative communication between patient and clinician in which knowledge, values, and preferences are shared and a process of common deliberation leads to a treatment decision. As the treatment decision for low-risk DTC is highly preference sensitive, SDM is even more relevant in thyroid cancer care to ensure that decisions made are consistent with each patient's preference. However, it can be difficult to achieve in standard clinical encounters because of the clinician's inability to establish patient values as well as patient's limited knowledge, unrealistic outcome expectations, and decisional conflict. As evidenced by a systematic review on the decision-making process in thyroid cancer management, many clinicians expressed difficulty in performing SDM as due to concerns with overwhelming patients with detailed information regarding disease and treatment options and struggled to find the right question to elicit patients' preference and value. Instead, the clinicians tailored treatment recommendation based on their perception of patient's level of fear, anxiety and risk tolerance, often without explicit discussion of patient's feelings. As a result, clinicians may be at risk of making recommendations biased by their own beliefs and values and the treatment received may not reflect patients' actual treatment goals.

Patient decision aids (PDA) are condition-specific decision-making tools that facilitate SDM by providing plain-language information about the potential risks (short- and long-term side effects), benefits, and uncertainties related to treatment, and information on how QoL and daily life could be affected. PDAs also help patients to clarify their values regarding options. PDAs can be in the format of web-page, pamphlet or video. Whilst PDAs have been developed for other cancers and diseases such as prostate cancer, breast cancer, diabetes mellitus and rheumatoid arthritis, to date there is no PDA for low-risk DTC. The investigators have developed a PDA for adult patients with low-risk DTC. Use of a PDA in low-risk DTC should increase patient's health knowledge, reduce uncertainty about which decision to make (decision conflict), improve decisional satisfaction, improve accuracy of risk perception of the outcome and help patient to make choices better matched to their personal values. In the long-term this will decrease patient's anxiety and distress, improve their physical and emotional functioning and their overall health related QOL.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18
* Both genders
* Patients who are diagnosed of low-risk well-differentiated thyroid carcinoma (papillary thyroid carcinoma or follicular carcinoma) with size of 1-4cm. This is either:

  1. Diagnosed pre-operatively by fine-needle aspiration cytology (FNAC) with Thy5 grade [see appendix for the Thy classification] or
  2. Confirmed following diagnostic hemithyroidectomy
* Able to communicate in spoken and written English

Exclusion Criteria:

* Patients who are diagnosed with thyroid cancer with adverse features (i.e. poor differentiated cytology or tall cell, columnar cell, Hurthle cell, and solid variant cytology)
* Patients who are diagnosed with thyroid cancer which is multifocal, bilateral, with extrathyroidal extension, with perineural invasion or angioinvasion.
* Patients who are diagnosed with thyroid cancer with clinically or radiologically involved nodes or distant metastases
* Patients who are diagnosed with thyroid cancer which is of a familial disease
* Patient who is either Pregnant or breast-feeding
* Patient with hyper- or hypothyroidism who is a candidate for surgery
* Patient who is concurrently diagnosed with any medullary, anaplastic, lymphoma, or parathyroid disease
* Patients who had previous thyroidectomy for reasons other than diagnostic hemithyroidectomy for their recent cancer diagnosis.
* Patients who are cognitively impaired or have a mental health condition and are therefore unable to give consent
* Patient who is not able to read write and speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be identified from the Thyroid MDT lists at the respective study centres by the local head and neck surgical team (patient's direct care team)
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-14 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | From enrolment for 9 months
  Successful recruitment rate of all eligible patients: the percentage of eligible patients who agree to participate out of all eligible patients screened and its 95% confidence interval.

SECONDARY OUTCOMES:
Percentage of participants in PDA arm who use the PDA-TC | From enrolment for 9 months
  Percentage of participants in PDA arm who use the PDA-TC to assist with the decision making process for their cancer treatment.
Difference of the overall score of the decisional conflict scale | From enrolment for 9 months
  The difference of the overall score of the decisional conflict scale after the consultation with and without the use of PDA-TC. The decisional conflict scale is a 5-point scale with 16 items and the lower the score, the better the outcome. This questionnaire is completed after the initial and second consultation. The satisfaction with decision scale is a 5-point scale with 6 items and the higher the score, the better the outcome. This questionnaire is completed after the second consultation. The preparation for decision making scale is a 5-point scale with 10 items and the higher the score, the better the outcome. The questionnaire is taken after the second consultation.

CONTACTS AND LOCATIONS:
Locations (1):
- Wrightington, Wigan and Leigh Teaching Hospitals NHS Foundation Trust, Wigan, United Kingdom